CLINICAL TRIAL: NCT05212766
Title: Role of the Oral Microbiome & Mucosal Immunity in COVID-19 Disease: Diagnostic/Prognostic Utility in South Asian Populations
Brief Title: Role of the Oral Microbiome & Mucosal Immunity in COVID-19 Disease
Acronym: MIMSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); UK Research and Innovation (Other)
Responsible Party: Sponsor
Other Study IDs: MIMSA
Record Dates: First submitted 2022-01-24; First posted 2022-01-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: COVID-19; Microbial Colonization; Oral Disease; Periodontal Diseases; Innate Inflammatory Response; Mucosal Infection
Keywords: COVID-19; periodontal disease; oral health; mucosal immunity
MeSH Terms: conditions — COVID-19; Communicable Diseases; Mouth Diseases; Periodontal Diseases; Inflammation | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Whole mouth fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Vaccinated or unvaccinated uninfected South Asian ethnicity: Participants will have not experienced infection (positive test) - we will aim to recruit both vaccinated and unvaccinated individuals although the latter may be harder to recruit. They will identify as of South Asian ethnicity. Uninfected subjects, will be recruited by advertisement within KCL or social media, from non-COVID in-patients or outpatients or attending A&E at GSTT and at SARS-CoV2 antigen testing centres and vaccination centres and at PIC sites.
  Interventions: Biological: COVID vaccination; Diagnostic Test: Oral examination
- Asymptomatic / mild infected South Asian ethnicity: Participants will have experienced asymptomatic or mild infection (positive test). They will identify as of South Asian ethnicity. Volunteers or subjects attending SARS-CoV2 testing centres who are found to be antigen positive or In-patients who have positive Covid tests and designated as asymptomatic/mild but admitted for non-covid reasons or those attending A&E with COVID but designated as mild/asymptomatic
  Interventions: Biological: COVID infection; Biological: COVID vaccination; Diagnostic Test: Oral examination
- Symptomatic infected South Asian ethnicity: Participants will have experienced moderate or severe symptomatic infection (positive test, admission). They will identify as of South Asian ethnicity. Patients either seen at GSTT or admitted as in-patients to GSTT or KCH and found to be SARS-CoV2 positive by RT-PCR in nasopharyngeal samples and designated as moderate/severe on the NIH/NIMR COVID severity scale.
  Interventions: Biological: COVID infection; Biological: COVID vaccination; Diagnostic Test: Oral examination
- Infected recovered South Asian ethnicity: Participants will have experienced moderate or severe symptomatic infection (positive test, admission) and recovered. They will identify as of South Asian ethnicity.
  Interventions: Biological: COVID infection; Biological: COVID vaccination; Diagnostic Test: Oral examination
- Vaccinated or unvaccinated uninfected Caucasian ethnicity: Participants will have not experienced infection (positive test) - we will aim to recruit both vaccinated and unvaccinated individuals although the latter may be harder to recruit. They will identify as of Caucasian ethnicity. Uninfected subjects, will be recruited by advertisement within KCL or social media, from non-COVID in-patients or outpatients or attending A&E at GSTT and at SARS-CoV2 antigen testing centres and vaccination centres and at PIC sites.
  Interventions: Biological: COVID infection; Biological: COVID vaccination; Diagnostic Test: Oral examination
- Asymptomatic / mild infected Caucasian ethnicity: Participants will have experienced asymptomatic or mild infection (positive test). They will identify as of Caucasian ethnicity. Volunteers or subjects attending SARS-CoV2 testing centres who are found to be antigen positive or In-patients who have positive Covid tests and designated as asymptomatic/mild but admitted for non-covid reasons or those attending A&E with COVID but designated as mild/asymptomatic
  Interventions: Biological: COVID infection; Biological: COVID vaccination; Diagnostic Test: Oral examination
- Symptomatic infected Caucasian ethnicity: Participants will have experienced moderate or severe symptomatic infection (positive test, admission). They will identify as of Caucasian ethnicity. Patients either seen at GSTT or admitted as in-patients to GSTT or KCH and found to be SARS-CoV2 positive by RT-PCR in nasopharyngeal samples and designated as moderate/severe on the NIH/NIMR COVID severity scale.
  Interventions: Biological: COVID infection; Biological: COVID vaccination; Diagnostic Test: Oral examination
- Infected recovered Caucasian ethnicity: Participants will have experienced moderate or severe symptomatic infection (positive test, admission) and recovered. They will identify as of Caucasian ethnicity
  Interventions: Biological: COVID infection; Biological: COVID vaccination; Diagnostic Test: Oral examination

INTERVENTIONS:
Biological: COVID infection — Infections with COVID 19
  Groups: Asymptomatic / mild infected Caucasian ethnicity; Asymptomatic / mild infected South Asian ethnicity; Infected recovered Caucasian ethnicity; Infected recovered South Asian ethnicity; Symptomatic infected Caucasian ethnicity; Symptomatic infected South Asian ethnicity; Vaccinated or unvaccinated uninfected Caucasian ethnicity
Biological: COVID vaccination — Vaccination against COVID 19
Diagnostic Test: Oral examination — Assessment of oral and periodontal health status

SUMMARY:
Determining whether in the mouth there are differences between the participant groups in the nature and activity of mucosal innate immunity, in immune responses to SARS-COV2 antigens, or in the oral microbiome

DETAILED DESCRIPTION:
Cross sectional with longitudinal component

* Stimulated whole mouth fluid (SWMF) and blood samples from South Asian and non-Asian populations
* Controls, and COVID-19 patients in both populations.
* Oral disease questionnaire and clinical examination
* Separation of SWMF into pellet for DNA extraction for microbiomics and supernatant for cell phenotype analysis, cytokines and antibodies to SARS-CoV2 antigens

ELIGIBILITY:
Inclusion Criteria:

* • South Asian and White British persons and those diagnosed with symptomatic or asymptomatic COVID-19 infection.

  * Aged 18 or over. Able to understand and consent.
  * Uninfected subjects: no history of COVID-19; not vaccinated; (negative for anti-SARS-CoV2 nucleoprotein antibodies at lab)
  * For patient groups: Confirmed COVID-19 positivity, symptoms and symptom onset within the past 21 days; Be recently hospitalised with COVID-19 disease; Have COVID-19 disease proven by PCR testing for SARS-CoV-2 within the last 21 days; COVID disease severity graded as per NIH/WHO.
  * Recovered groups: Have had COVID-19 disease proven by PCR testing for SARS-CoV-2. COVID disease severity graded as per WHO or NIH equivalent criteria
  * Those willing to participate on a single occasion but unwilling to participate with longitudinal samples will not be excluded.
  * Smoking, obesity, diabetes, heart disease, antibiotics or treatment related to COVID is not excluded.

Exclusion Criteria:

* • Those patients unwilling to participate, those unable to understand sufficiently to give informed consent and those unable to participate due to the severity of COVID-19 disease. Those patients classified as not either South Asian or White British heritage.

  * Patients with malignancy, pregnancy, long term immune suppression, inability to give informed consent, not willing or able to have oral examination.
  * Diabetes not excluded but screening for diabetes will be performed: glucose will be assessed in blood/serum sample (150ul).

Exclusion criteria summary:

* Critically ill participants who cannot give informed consent
* Those who are not willing to have an oral examination, or donate blood or saliva samples.
* Those who cannot chew / drool to provide a SWMF sample due to severe/critical medical conditions
* Participants with known malignancies or who are pregnant
* Participants who are on long-term immunosuppressants (e.g. for autoimmune diseases)
* Participation in other current research that is designed to, or is expected to alter the immune response.
* Inability to communicate, understand or read English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants, both South Asian and White British will be recruited by advertisement within KCL or social media, from non-COVID in-patients or outpatients or attending A&E at GSTT and at SARS-CoV2 antigen testing centres and vaccination centres and at PIC sites. Also patients either seen at GSTT or admitted as in-patients to GSTT or KCH and found to be SARS-CoV2 positive. Patients who have had COVID may be invited directly to participate by advertising at sites specified above or be attending either the post-COVID or ICU follow-up outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between oral mucosal immunity and microbiome on COVID outcomes in different ethnic groups | 16 weeks
  Multiple assessments

SECONDARY OUTCOMES:
Impact of immunity and oral microbiome | 16 weeks
  To determine whether the presence of pre-existing oral disease is related to susceptibility to SARS-CoV2 infection, to severity of COVID-19 disease or relates to the nature of mucosal immunity and to the composition and activity of the oral microbiome
Impact of pre-existing oral disease | 16 weeks
  To determine whether the presence of pre-existing oral disease is related to susceptibility to SARS-CoV2 infection, to severity of COVID-19 disease or relates to the nature of mucosal immunity and to the composition and activity of the oral microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Challacombe, PhD, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Trust / King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
It is likely that anonymised data may be shared with colleagues carrying out a linked study in India, although the exact nature of this yet to be confirmed